CLINICAL TRIAL: NCT07229079
Title: The Effectiveness of Basic Body Awareness Therapy Combined With Short Foot Exercises in Individuals With Pes Planus
Brief Title: The Effectiveness of Basic Body Awareness Therapy in Individuals With Pes Planus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, Fatma Betül YARDIMCI, RESEARCH ASSISTANT, Mardin Artuklu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FBYDRTEZ
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pes Planus
Keywords: Short Foot Exercises (SFE); Basic Body Awareness Therapy (BBAT); Pes Planus; Balance; Proprioception; Flatfoot
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the Control Group (Short Foot Exercises only) or the Experimental Group (BBAT + SFE) in parallel arms for comparison.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BBAT Group (Experimental): Participants will receive Short Foot Exercises (SFE) plus Basic Body Awareness Therapy (BBAT).
  Interventions: Behavioral: Basic Body Awareness Therapy (BBAT); Behavioral: Short Foot Exercises (SFE)
- Control Group (Active Comparator): Participants will receive only Short Foot Exercises (SFE).
  Interventions: Behavioral: Short Foot Exercises (SFE)

INTERVENTIONS:
Behavioral: Basic Body Awareness Therapy (BBAT) — Participants will perform Basic Body Awareness Therapy (BBAT) combined with SFE for 8 weeks. BBAT sessions are 45 minutes, twice weekly in small groups under a certified physiotherapist. Exercises target postural control, motor coordination, body awareness, balance, and functional movement, progressing from supine to sitting, standing, and walking positions. After each BBAT session, participants perform SFE following the same progression as the Control Group.
  Arms: BBAT Group
Behavioral: Short Foot Exercises (SFE) — Participants will perform Short Foot Exercises (SFE) for 8 weeks. Sessions are twice weekly under physiotherapist supervision in small groups (3-8 participants) and 5 days/week at home. Exercises progress from sitting (weeks 1-2), standing (weeks 3-4), single-leg (weeks 5-6), to functional activities (weeks 7-8). Each session lasts ~20 minutes, 3 sets of 10 reps with 1-minute rest. Participants receive instruction on proper technique and adherence is monitored online

SUMMARY:
This study investigates whether adding Basic Body Awareness Therapy (BBAT) to Short Foot Exercises (SFE) improves pes planus, balance, and body awareness in adults with flexible pes planus. Fifty participants aged 18-45 will be randomly assigned to either a BBAT + SFE group or an SFE-only control group. The interventions will last eight weeks with supervised sessions twice weekly and additional home exercises. Outcomes will be measured before, after, and two months post-intervention.

DETAILED DESCRIPTION:
Pes planus is a common orthopedic condition characterized by the collapse of the medial longitudinal arch of the foot, which negatively affects lower extremity biomechanics, postural stability, and balance. Currently, interventions targeting muscle activation-such as short foot exercises (SFE)-are widely used in the management of pes planus. However, it is believed that holistic approaches incorporating sensory input and body awareness may further enhance functional outcomes in these individuals. Basic Body Awareness Therapy (BBAT) is a physiotherapeutic method designed to improve movement quality, balance, and posture. In this study, BBAT will be applied for the first time in individuals with pes planus. This project aims to investigate the effects of BBAT, when combined with SFE, on medial longitudinal arch height, foot function, gait, balance, proprioception, plantar sensation, and body awareness in individuals with pes planus. The study will be conducted as a randomized controlled trial. Fifty participants who meet the inclusion criteria will be randomly assigned into two groups of 25: a BBAT group (SFE + BBAT) and a control group (SFE only). Interventions will be administered twice a week for a duration of eight weeks. Assessments will be conducted at three time points: before the intervention, immediately after the eight-week intervention period, and two months post-intervention (follow-up). This study aims to demonstrate that BBAT can provide significant improvements in both somatic and sensory parameters in individuals with pes planus, offering a holistic complement to traditional exercise-based approaches. In doing so, it is expected to contribute an innovative perspective to clinical physiotherapy practices and address a significant gap in the existing literature.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years
* Willing to participate in the study
* Flexible pes planus (Navicular Drop ≥10 mm and positive Jack's Toe Raise Test)

Exclusion Criteria:

* Pain in lower extremity joints
* Obesity (BMI >30)
* Pregnancy
* Systemic, neuromuscular, or neurological disorders
* Posterior tibial tendon dysfunction (unable to perform heel-rise test)
* History of lower limb surgery
* Previous treatment for pes planus or use of foot orthoses
* Lower extremity injury in past 6 months
* Orthopedic conditions other than pes planus and mild hallux valgus (Manchester Scale C or D excluded)
* Participation in regular exercise program in past 6 months
* Prior personal experience with TBFT and/or short foot exercises

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Navicular Drop Test | Baseline (pre-intervention), post-intervention (8 weeks), follow-up (2 months after intervention)
  Assessment of medial longitudinal arch height to determine presence and severity of pes planus. Test performed in both sitting (non-weight-bearing) and standing (weight-bearing) positions. Difference ≥10 mm indicates pes planus.
Dynamic Balance | Baseline, post-intervention (8 weeks), follow-up (2 months)
  Y Balance Test measuring reach distance in anterior, posteromedial, and posterolateral directions. Results normalized to leg length.
Proprioception | Baseline, post-intervention (8 weeks), follow-up (2 months)
  Active and passive joint position sense of the ankle measured with digital goniometer. Eyes closed; angular error from target angle recorded.
Light Touch Sensation | Baseline, post-intervention (8 weeks), follow-up (2 months)
  Semmes-Weinstein Monofilament Test at seven foot reference points. Threshold of sensation recorded.

SECONDARY OUTCOMES:
Foot Function Index - Pain Subscale | Baseline, post-intervention (8 weeks), follow-up (2 months)
  The Pain subscale of the Foot Function Index (FFI) assesses foot pain during daily activities. It includes 9 items rated on a 0-10 Likert-type scale. Higher scores indicate worse pain.self-rate 23 items using a visual analog scale.
Foot Function Index - Disability Subscale | Baseline, post-intervention (8 weeks), follow-up (2 months)
  The Disability subscale of the Foot Function Index (FFI) evaluates difficulty in performing functional activities. It contains 9 items scored on a 0-10 Likert-type scale. Higher scores indicate greater disability.
Foot Function Index - Activity Limitation Subscale | Baseline, post-intervention (8 weeks), follow-up (2 months)
  The Activity Limitation subscale of the Foot Function Index (FFI) measures limitations in essential daily activities. It consists of 5 items rated on a 0-10 Likert-type scale. Higher scores indicate greater activity limitation.
Foot Function Index - Total Score | Baseline, post-intervention (8 weeks), follow-up (2 months)
  The Total Score of the Foot Function Index (FFI) is calculated by combining all pain, disability, and activity limitation items (23 items in total). Each item is rated on a 0-10 Likert-type scale. The total score reflects the overall foot-related functional status, with higher scores indicating worse function.
Static Balance | Baseline, post-intervention (8 weeks), follow-up (2 months)
  Flamingo Balance Test. Participant stands on one leg on a narrow beam for 1 minute; balance errors recorded.
Gait Performance | Baseline, post-intervention (8 weeks), follow-up (2 months)
  10-Meter Walk Test performed at comfortable walking speed. Time recorded and averaged over three trials.
Body Awareness | Baseline, post-intervention (8 weeks), follow-up (2 months)
  Body Awareness Questionnaire assessing participant's perception of bodily sensations and processes. Score range 18-126; higher scores indicate better awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Betül Yardımcı, MSc, Principal Investigator — Mardin Artuklu University
Locations (1):
- Mardin Artuklu University, Mardin, Mardi̇n, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No